CLINICAL TRIAL: NCT04835077
Title: Comparison of the Effectiveness of Structured Aerobic Exercises and Postural Stabilization Exercises in Patients With Fibromyalgia Syndrome
Brief Title: Aerobic Exercises and Postural Stabilization Exercises in Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mustafa Yilmaz, MSc Physiotherapsit, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulC
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia Syndrome; Physiotherapy; Rehabilitation
Keywords: Aerobic Exercise; Postural Control; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Control Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Aerobic Exercises (Experimental): Following the training on aerobic exercise content and effectiveness;
  1. First Week; participants 5 minutes warm-up, 20 minutes of aerobic exercise with 60-70% of maximum heart rate, and 5 minutes of cool down.
  2. In the following weeks, the aerobic exercise duration of all participants will be increased by 5 minutes compared to the previous week.
  3. The duration of the sessions in the 7th and 8th weeks will progressively progress to 40 minutes and the intensity to 75-80% of the maximum heart rate.
  Interventions: Other: aerobic exercise
- Postural Stabilization Exercises (Experimental): Exercises; It will consist of postural exercises to be done in prone, supine, side lying, crawling, sitting and standing positions. All exercises will be done in 2 sets per day, the number of repetitions will be determined individually and progressed.
  1. Breathing exercises
  2. Four-way stretching and strengthening of the neck muscles
  3. Shoulder girdle stretching and strengthening exercises
  4. Hip flexors, hamstring, itb, lumbar extensor stretching and strengthening
  5. Lying down exercises in the crawling position
  6. Shuttle movement
  7. Plank movement
  8. Toe taps
  9. Bridging
  10. Straight leg lift
  11. Straight leg raises in side-lying
  12. Prone knee flexion
  Interventions: Other: postural stabilization exercises
- Control (No Intervention): The individuals without any treatment will continue their normal lives and will be included in the study as a control group. Exercise will be given after 8 weeks.

INTERVENTIONS:
Other: aerobic exercise — Structured aerobic exercises (Each session will consist of 50 minutes and will be divided into three parts: 5 minutes of warm-up exercises, 40 minutes of aerobic exercises, 5 minutes of cool down exercises) will be taught in the first session.
  Arms: Structured Aerobic Exercises
Other: postural stabilization exercises — Structured postural stabilization exercises (strengthening exercises, balance-coordination exercises, flexibility exercises) will be taught in the first session.
  Arms: Postural Stabilization Exercises

SUMMARY:
Fibromyalgia Syndrome (FMS) is a chronic rheumatic disease characterized by a wide range of symptoms such as widespread muscle pain, fatigue, sleep disturbances, anxiety-depression, impaired balance, falling risk, poor physical condition, cognitive dysfunction, and irritable bowel syndrome.

The aim of the study; It is a comparison of the effectiveness of aerobic exercises and postural stabilization exercises that are structured to reduce the pain severity, fatigue, sleep problems and anxiety-depression levels of patients who are being followed up with a diagnosis of FMS, and to increase the duration of physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 25-60 According to the 2013 American College of Rheumatology (ACR) diagnostic criteria, the Pain Placement Score (AES) is 17 and the Symptomatic Effect Score (SES) is ≥21.
* FMS symptoms persist for more than 3 months
* Ability to adapt to exercise
* Having the ability to use the necessary devices for web-based training

Exclusion Criteria:

* Any disease that may hinder exercise
* Finding cardiological problems for aerobic exercises
* Presence of loss of sense and sense of position
* Presence of an unhealed fracture or surgical wound Patients with mental / psychotic disorders

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | change from baseline at 8 weeks
  This scale; It measures 10 different characteristics: physical function, feeling unwell, not going to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Except for the sense of well-being, lower scores indicate improvement or less affected by the disease. FIQ is filled by the patient. The maximum possible score for each subtitle is 10. Thus, the total maximum score is 100. While the average FM patient gets 50 points, more severely affected FM patients usually score above 70.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | change from baseline at 8 weeks
  VAS; It is a scale that provides a one-dimensional measurement of pain intensity in different adult populations. It usually consists of a 10 cm long horizontal (HVAS) or vertical (VVAS) line. In measuring the severity of pain; A score of 0 is defined as no pain, a score of 10 as worst pain possible or worst imaginable pain. Although the period of time when pain is questioned varies, the most common time for the patient's pain is the current pain or the pain experienced in the last 24 hours.

OTHER OUTCOMES:
Brief Pain Inventory (BPI) | change from baseline at 8 weeks
  The BPI questionnaire is a short, easy-to-apply assessment method that can be used to assess pain. It includes simple 0 to 10 numerical evaluation scales that are easy to understand and translate into different languages. In the short pain inventory, a score of 1-4 of the worst pain is defined as mild pain, 5-6 as moderate pain, and 7-10 as severe pain. Evaluates the severity of pain, localization of pain, medical treatments for pain, and the effect of pain on daily functions, and questions how much pain has been reduced in the last 24 hours or last week. It takes a short time, like 5-10 minutes, to answer all questions.
Pittsburgh Sleep Quality Index (PSQI) | change from baseline at 8 weeks
  PSQI is a 19-item self-report scale that evaluates sleep quality and disorder over the past month. Each item of the test is equally scored between 0 and 3. The scale consists of 7 subscales that evaluate subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping pills and daytime functionality loss. The total PSQI score ranging from 0 to 21 is obtained by summing the subscales. A total PSQI score greater than 5 indicates that the individual's sleep quality is insufficient with 89.6% sensitivity and 86.5% specificity, and indicates severe impairment in at least two areas, or moderate deterioration in three areas.
Fatigue Severity Scale (FSS) | change from baseline at 8 weeks
  The person indicates how much they agree with each item by choosing numbers from 1 to 7. 1 indicates that they disagree at all, 7 indicates that they agree completely. The score range of the scale, which consists of 9 questions in total, is 9-63. A score of 36 or higher indicates severe fatigue. The total score is calculated by taking the average of 9 items. The cut-off value for pathological fatigue was set at 4 and above. The lower the total score, the less fatigue.
2 Minute Walking Test | change from baseline at 8 weeks
  Subjects begin to walk for 2 minutes at their own walking pace in the 21-meter corridor marked from the starting line, wearing their shoes and using their normal walking aids. The lines at both ends of the floor of the corridor indicate where the subjects will turn. The evaluator walks behind the subjects to ensure their safety and to minimize changes in pacing speed while walking. It also keeps time using a digital stopwatch.
Short Form Health Survey (SF-36) | change from baseline at 8 weeks
  It is one of the most common generic measures used to measure quality of life. This scale examines 8 dimensions of health such as physical function, role restrictions, social function, mental health, energy, pain and general perception of health with 36 items. The scale gives a separate total score for each subscale rather than just a single total score, and the scores range from 0 to 100. While 100 points indicate good health, 0 points indicate poor health.
International Physical Activity Questionnaire Short Form (IPAQ Short Form) | change from baseline at 8 weeks
  IPAQ Short Form; It consists of nine questions measuring the intensity of physical activity. The questions provide information about physical activities (climbing stairs, walking, shopping, sitting time) in the last 7 days. From these data, the total weekly physical activity level (MET / hour / week) is classified as low, medium and high. Individuals who indicate that they do not have physical activity must have a low physical activity level x ≤ 600 MET / minute / week, and in order to be at an intense or moderate level of physical activity, total physical activity must be attained to a minimum of x ≥ 600-3000 MET / minute / week.
PostureZone Mobile Application | change from baseline at 8 weeks
  PostureZone mobile application is a new application that makes posture assessment more effective in different environments. Free versions of this easy-to-use and fast application are available on mobile devices. For posture analysis, participants are photographed anteriorly and laterally in front of a flat surface using the device camera. Then, after manually marking the anatomical points on the photograph, the program performs the analysis. With this program, shift and tilt values occurring in the head, shoulder, rib and hip in the anterior and shift and tilt values occurring in the head, shoulder, hip and knee in the lateral can be calculated. If desired, the total shift and tilt values obtained from both angles can be saved. This program, which aims to obtain reliable information through the processing and interpretation of photographic images, can be used in postural assessments thanks to the quantification of linear and angular measurements.
Plank position time | change from baseline at 8 weeks
  Plank; It is called a type of exercise that develops the leg and chest muscles, especially the abdominal muscles, and is done 45 degrees with the ground. Plank movement improves bodily qualities such as strength, balance and endurance when properly applied. This movement works the entire abdominal muscle. Apart from that, it strengthens the neck, back, waist, chest and front / back leg muscles; Corrects posture disorders. It ensures that the shoulders are back and the breasts are high. The whole body is tightened with the help of the fingertip on the elbows and the head is facing forward. The evaluator keeps time using a digital stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA YILMAZ, Principal Investigator — MSc Physiotherapist
Locations (1):
- Mustafa Yilmaz, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Walker J. Fibromyalgia: clinical features, diagnosis and management. Nurs Stand. 2016 Sep 28;31(5):51-63. doi: 10.7748/ns.2016.e10550. PMID 27682568
- [Background] Vincent A, Lahr BD, Wolfe F, Clauw DJ, Whipple MO, Oh TH, Barton DL, St Sauver J. Prevalence of fibromyalgia: a population-based study in Olmsted County, Minnesota, utilizing the Rochester Epidemiology Project. Arthritis Care Res (Hoboken). 2013 May;65(5):786-92. doi: 10.1002/acr.21896. PMID 23203795
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367